CLINICAL TRIAL: NCT06138548
Title: Bio-Integrative, Fiber-Reinforced Kneebar for Treating Subchondral Insufficiency of the Knee
Status: Enrolling by invitation | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Seth Sherman, Associate Professor, Stanford University
Other Study IDs: 72105
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Subchondral Insufficiency Fracture
Keywords: Ossio; Kneebar; Fracture; Subchondral insufficiency; Tibial overload; Femoral Overload
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subchondral Insufficiency: Those who have subchondral insufficiency with tibial or femoral overload in the knee and are receiving the TFNs as standard of care.
  Interventions: Device: Ossiofiber® Trimmable Fixation Nail

INTERVENTIONS:
Device: Ossiofiber® Trimmable Fixation Nail — OSSIOfiber® Trimmable Fixation Nails are equally strong in the initial stability and fixation strength - and superior in rotational resistance to traditional metal cannulated headless compression screws.*

SUMMARY:
The OSSIOfiber® Trimmable Fixation Nails are indicated for maintenance of alignment and fixation of bone fractures, osteotomies, arthrodesis and bone grafts in the presence of appropriate additional immobilization (e.g., rigid fixation implants, cast, brace). The hypothesis is that the use of OSSIOfiber® Trimmable Fixation Nails for treating subchondral insufficiency of the knee will result in improvement of patient-reported outcomes and imaging findings. The primary objective of this study is to evaluate the effectiveness of implanting bio-integrative OSSIOfiber® Trimmable Fixation Nails, organized in a bi-cortical rafter formation within the tibia or femur for the management of subchondral insufficiency. This use is not considered off-label because the TFNs are being used in the way they are intended to be used via FDA approval.

ELIGIBILITY:
Inclusion Criteria:

1. Has had knee pain in study knee lasting at least 3 months
2. Candidate for knee arthroscopy due to meniscal tear, loose body, unstable articular cartilage or mechanical symptoms.

Exclusion Criteria:

1. Current tobacco use or has quit within 3 months of study enrolment.
2. Substance abuse history.
3. Diabetes mellitus, HbA1c>8
4. High surgical risk due to pre-existing conditions.
5. Currently pregnant or has plans to become pregnant prior to surgery.
6. Active infection or history of chronic infection in study knee.
7. Will require concomitant procedures within study knee, including but not limited to ligament reconstruction, tendon repair, meniscus repair, microfracture, osteotomy, or osteochondral transplantation. (Meniscal tears, including chronic, are acceptable if no repair is required)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those who have subchondral insufficiency of the knee with tibial or femoral overload.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | 3 months post-operatively
  The overall KOOS score combines pain and function domains. KOOS is out 100, where 0 equates to extreme pain and 100 equates to no pain.
Knee injury and Osteoarthritis Outcome Scale Score (KOOS) | 6 months post-operatively
  The overall KOOS score combines pain and function domains. KOOS is out 100, where 0 equates to extreme pain and 100 equates to no pain.

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR.) | 6 months post-operatively
  Measures the knee health of individuals following surgery
International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form | 6 months post-operatively
  IKDC measures: symptoms, athletic activity, and knee function.
Veterans Rand-12 (VR-12) Health Survey Scale Score | 6 months post-operatively
  VR-12 combines measures of general health perceptions, physical functioning, role limitations due to physical and emotional problems, bodily pain, fatigue , social functioning, and mental health
Numeric Pain Reported Scale Score | 6 months post-operatively
  Measures a subject's perceived pain level. This score is usually on a scale of 0-10 with 0 equating to no pain and 10 equating to the worst pain imaginable.
PROMIS Pain Interference Score | 6 months post-operatively
  Measures what level pain hinders a patient's engagement in several activities including social, cognitive, physical, and recreational activities. There are 7 sub items and each are rated from a scale of 0-10 where 0 means it does not interfere and 10 means it completely interferes. These contribute to a final score ranging anywhere from 0-70.
PROMIS Depression Score | 6 months post-operatively
  Measures self-reported negative mood (sadness, guilt), views of self (self- criticism, worthlessness), and social cognition (loneliness, interpersonal alienation), as well as decreased positive affect and engagement (loss of interest, meaning, and purpose). Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40. Higher scores indicate greater severity of depression.
PROMIS Physical Function Score | 6 months post-operatively
  Measures the level of physical function for patients with a wide variety of impairments that may limit the patient's physical capability. This score is on a scale from 0-100 with 0 equating to no physical function and 100 equating to optimal physical function.
Incidence Assessments | Up to 24 month post-operatively.
  Assessment of the incidence of re-operations, revision surgeries, or additional management of the study knee outside of postoperative rehabilitation.
Degree of knee ligament healing | 6, 12, and 24 months
  To see how the knee ligament is healing by MRI assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Seth L Sherman, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - Rush University, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No